CLINICAL TRIAL: NCT01353326
Title: Randomized Clinical Trial of a Cemented Versus Cementless Femoral Component for Metal on Metal Hip Resurfacing Assessing Bone Mineral Density
Brief Title: Bone Mineral Density (BMD) in Cemented Versus Cementless Hip Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Corin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008058-01H
Record Dates: First submitted 2009-09-30; First posted 2011-05-13 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
Keywords: non-inflammatory degenerative joint disease; hip resurfacing; bone mineral density; cemented; cementless
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cementless Hip Resurfacing (Active Comparator): Patients randomized into the Cementless Hip Resurfacing Group will have their hip resurfaced with the cementless Cormet / Corin Hip Resurfacing System.
  Interventions: Device: Cormet
- Cemented Hip Resurfacing (Active Comparator): Patients randomized into the Cemented Hip Resurfacing Group will have their hip resurfaced with the cemented Conserve Plus Total Resurfacing Hip System.
  Interventions: Device: Conserve

INTERVENTIONS:
Device: Cormet — Cementless hip resurfacing system
  Other Names: Cormet Hip Resurfacing System; Corin
  Arms: Cementless Hip Resurfacing
Device: Conserve — Cemented hip resurfacing system
  Other Names: Conserve Plus Total Resurfacing Hip System; Wright
  Arms: Cemented Hip Resurfacing

SUMMARY:
The purpose of this study is to compare the bone mineral density of patients who have undergone either cemented or cementless hip resurfacing.

DETAILED DESCRIPTION:
Recent research is inconclusive regarding the degree to which the density or strength of the bone around the hip implant is preserved following a hip resurfacing system. Certainly, there are many factors which contribute to the preservation of bone mineral density - we are studying the role of cement. More specifically, we are trying to compare outcomes between patients who receive the cementless Cormet Hip Resurfacing System to those who receive the cemented CONSERVE® Plus Total Resurfacing Hip System. Therefore, the primary purpose of the current study is to compare the bone mineral density between the cementless and cemented hip resurfacing systems. We are also comparing patients who receive these two different hip systems in terms of their x-rays and how they are managing with their hip.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing primary hip surgery for Noninflammatory Degenerative Joint Disease
* must be skeletally mature, as determined by Risser sign or reaching 18 years of age
* Is reasonable expectation that patient will remain available for all FU's scheduled over course of 5 years

Exclusion Criteria:

* Previous fusions, acute femoral neck fractures, and above knee amputations
* evidence of active local infection
* neurologic or musculoskeletal disease that may adversely affect gait or weight bearing
* having previously undergone ipsilateral hemi resurfacing, total resurfacing, total bipolar, unipolar or total hip replacement device
* BMI >35
* neuropathic joints
* severe documented psychiatric disease
* patients requiring structural bone grafts
* documented allergy to cobalt chromium molybdenum
* ipsilateral girdlestone
* sickle cell disease
* significant femoral head or neck deformity, or significant acetabular wall deficiency
* patients with renal failure, defined as serum creatinine greater that 180 µmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05-15 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percent change in BMD (g/cm2) | 12 months
  The primary outcome is percent change in BMD (g/cm2) from baseline to the 1-year post-operative interval, as measured radiographically in zone L1. Analysis of periprosthetic BMD will be achieved using 6 zones of the femoral neck, which have been used in previous studies

SECONDARY OUTCOMES:
Implant Migration | 24 months
  Radiographs will be taken preoperatively and until 24 months post-operatively to assess for any cup loosening. Implant migration, both vertical and horizontal, will be measured on serial radiographs using the computer-assisted Ein Bild Röentgen Analyse (EBRA) software for cup migration.
Harris Hip Score (HHS) Questionnaire | 24 months
  The Harris Hip Score (HHS) is intended to evaluate various hip disabilities and methods of treatment. The HHS is comprised of 4 domains: pain, function, absence of deformity, and range of motion. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points). The total score is calculated by summing the scores for the 4 domains. The higher the HHS, the less dysfunction.
WOMAC Questionnaire to assess functionality | 24 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) consists of 24 items divided into 3 subscales: Pain (5 items), stiffness (2 items), and function (17 items). This questionnaire is self-administered using the 5-point Likert-type scale (none, mild, moderate, severe, extreme). These correspond to an ordinal scale of 0-4. The scores are summed (0-100), where higher scores are indicative of worse pain, stiffness, and functional limitations.
RAND-36 Item Health Survey | 24 months
  The RAND-36 Item Health Survey assesses patient health-related quality of life and consists of 8 health concepts: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (3 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). It also includes a single item that provides an indication of perceived change in health. Each item is scored on a 0 to 100 range, with a high score defined as a more favourable health state. Scores are averaged together to create the 8 scale scores.
UCLA Activity Score | 24 months
  The UCLA Activity Score will be used to assess the patients highest-rated activity, regardless of the frequency or intensity of participation. Patients are asked to select 1 out of 10 possible answers that best fit their current activity level (0-10). Low values are indicative of a sedentary lifestyle, while higher values are indicative of high impact activities.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Paul Beaule, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa General Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Tice A, Kim P, Dinh L, Ryu JJ, Beaule PE. A randomised controlled trial of cemented and cementless femoral components for metal-on-metal hip resurfacing: a bone mineral density study. Bone Joint J. 2015 Dec;97-B(12):1608-14. doi: 10.1302/0301-620X.97B12.36110. PMID 26637673